CLINICAL TRIAL: NCT06390644
Title: Effect of Periorbital Massage on Dry Eye Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/701
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Control Groups; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periorbital Massage Therapy (Experimental): Participants in this arm will receive periorbital massage therapy administered by a trained practitioner.
  Interventions: Diagnostic Test: Periorbital Massage Therapy
- Control Group (Standard Care) (Other): Participants in this arm will receive standard care for dry eye disease.
  Interventions: Other: Control Group (Standard Care)

INTERVENTIONS:
Diagnostic Test: Periorbital Massage Therapy — Participants in this arm will receive periorbital massage therapy administered by a trained practitioner. The massage technique will involve gentle circular motions around the eye sockets and brow bone area, aiming to improve eyelid and tear gland function.
  Arms: Periorbital Massage Therapy
Other: Control Group (Standard Care) — Participants in this arm will receive standard care for dry eye disease, which include artificial tears. They will not receive periorbital massage therapy."
  Arms: Control Group (Standard Care)

SUMMARY:
This randomized controlled trial aims to investigate the efficacy of periorbital massage therapy in alleviating symptoms and improving clinical outcomes in patients diagnosed with dry eye disease.

DETAILED DESCRIPTION:
Participants will be randomized into either a periorbital massage intervention group or a control group receiving standard care. The intervention group will receive gentle periorbital massage techniques, while the control group will receive conventional dry eye treatments. The primary outcome measure will be assessed using the Schirmer Strips and Ocular Surface Disease Index (OSDI) questionnaire. This study holds promise for providing insights into the potential benefits of periorbital massage therapy as a complementary approach for managing dry eye disease symptoms and enhancing patients' overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of dry eye (such as burning, dryness or foreign body sensation)
* Ocular signs of dry eye (such as tear film instability, reduced tear production or meibomian gland dysfunction)
* Patients having moderate and severe dry eye disease according to schirmer test Willing and able to comply with the study protocol

Exclusion Criteria:

* Active ocular infection
* Ocular surgery within past 3 months
* Use of contact lenses
* Use of systemic medications that can affect tear production or tear quality
* Pregnancy or lactation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Schirmer Strips | 12 Months
  Schirmer's test is used to determine whether the eye produces enough tears to keep it moist. The test is performed by placing filter paper inside the lower lid of the eye. After 5 minutes, the paper is removed and tested for its moisture content.

SECONDARY OUTCOMES:
OSDI Questionnaire | 12 Months
  The Ocular Surface Disease Index (OSDI) is a questionnaire that has been validated to discriminate between normal, mild to moderate, and severe dry eye disease as defined by the physician's assessment and a composite disease severity score

CONTACTS AND LOCATIONS:
Locations (1):
- Usman Saleem Hospital and Fouzia Maternity Home Address: Usman Saleem Hospital and Fouzia Maternity Home, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No